CLINICAL TRIAL: NCT05898048
Title: Cytomegalovirus Reactivation in Acute Necrotizing Pancreatitis
Brief Title: CMV Reactivation in Acute Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2023-51-DM-130
Record Dates: First submitted 2023-05-27; First posted 2023-06-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Necrotizing Pancreatitis
Keywords: Critically ill; Cytomegalovirus; Reactivation; Intensive care unit
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients with the diagnosis of acute necrotizing pancreatitis (ANP) present with a wide spectrum of severity. These patients frequently require intensive care management. According to the revised Atlanta classification (2012), acute pancreatitis is divided into distinct subtypes, based on the presence or absence of necrosis. The mortality rates for sterile necrosis though comparatively low (5%-10%), but superinfection of the necrotic pancreas and peri-pancreatic tissue/ fluid collections increases the mortality rate considerably (up to one-third). The most common organisms isolated from the infected pancreatic necrosum are gram-negative bacteria mainly Escherichia coli and Klebsiella pneumoniae followed by gram-positive bacteria; however, with the increased use of antibiotic therapies in the ICU, the incidence of pancreatic fungal infections is also on a rise. Traditionally, critically ill patients have been considered immunocompetent but the immunomodulatory effects of sepsis may lead to reactivation of dormant viral infections. In recent years, Cytomegalovirus (CMV) reactivation in critically ill patients has been recognized with as high as 71% incidence with associated higher mortality, organ failure rates, duration of mechanical ventilation, nosocomial infections, and ICU length of stay. CMV reactivation had been studied in various cohorts in the ICU population, such as acute respiratory distress syndrome (ARDS) and septic shock exhibiting their impact on mortality. However, currently, no study is available investigating the role of CMV reactivation in patients with acute necrotizing pancreatitis. Therefore, the investigators aimed to study the prevalence of CMV reactivation and its viral load kinetics in critically ill patients with acute necrotizing pancreatitis.

DETAILED DESCRIPTION:
Background and Rationale for the Study Acute pancreatitis is one of the frequently encountered systemic diseases presenting with a wide spectrum of presentation ranging from mild disease which has a better outcome compared to severe disease which usually leads to admission to the intensive care unit (ICU), and is associated with high mortality. According to the revised Atlanta classification (2012), acute pancreatitis is now divided into two distinct subtypes, necrotizing pancreatitis and interstitial edematous pancreatitis (IEP), based on the presence or absence of necrosis. In severe acute pancreatitis, inflammation leads to peri-pancreatic fluid collections of which four distinct subtypes are identified. Acute necrotic collections (ANC) and walled-off necrosis (WON) which occur in patients with necrotizing pancreatitis, contain variable amounts of fluid and necrotic debris which can either be sterile or infective. The mortality rates for sterile necrosis remain comparatively low (5%-10%), but superinfection of the necrotic pancreas and peri-pancreatic tissue/ fluid collections increases the mortality rate considerably (20%-30%).

The infected pancreatic necrosum when cultured, usually demonstrates mono-microbial flora in 60-87% of patients and poly-microbial flora in 13-40% of patients. The most common organisms isolated are gram-negative bacteria, mainly Escherichia coli and Klebsiella pneumonia followed by gram-positive bacteria. With the increased use of antibiotic therapies in the ICU the incidence of pancreatic fungal infections is also on the rise. Fungal pancreatic infections, predominantly caused by Candida species, have been identified in up to one-half with a longer hospital stay and a lower one-year survival than patients with bacterial pancreatic infections only.

Traditionally, critically ill patients have been considered immunocompetent but the presence of sepsis and its immunomodulatory effects may lead to reactivation of dormant viral infections. In recent years, Cytomegalovirus (CMV) reactivation in critically ill patients has been recognized with as high as 71% incidence. Sepsis due to its immunomodulatory effects may lead to the reactivation of CMV due to the release of pro-inflammatory cytokines such as TNF-alpha and IL-1beta which has the ability to activate several transcription factors contributing to CMV reactivation. Studies showed that CMV infection in critically ill patients was consistently associated with undetectable IFN-γ T cell responses within the first 2 days of admission to the ICU and that viral load was inversely related to IFN-γ T cell responses. Similar results were found in septic patients who display immune system paralysis, reduced Th1 cell function, increased IL-10 production (anti-inflammatory), and global lymphopenia affecting natural killer cells (NK) quantitatively and qualitatively related to their interferon production.

Studies have documented significantly higher organ failure rates and mortality in critically ill patients with CMV reactivation. In a systematic review to investigate the association between CMV reactivation and clinical outcomes in immunocompetent critically ill patients, including Itwenty-two studies, CMV reactivation was associated with increased ICU mortality, overall mortality, duration of mechanical ventilation, nosocomial infections, and ICU length of stay. CMV reactivation has also been studied in specific critically ill cohorts, exhibiting their impact on mortality. The effect of CMV reactivation on mortality in immunocompetent acute respiratory distress syndrome (ARDS) patients has also been studied. Of 399 ARDS patients, 68 % were CMV seropositive and reactivation occurred in 27 % of them which was associated with overall increased ICU mortality. In another study among the septic shock cohort (329 patients), herpesvirus reactivations were documented in 68% of patients without prior immunodeficiency, and concluded that reactivations could be independently associated with mortality.

However, no studies are currently available investigating CMV reactivation in patients with acute necrotizing pancreatitis (ANP). The investigators aimed to study the prevalence of CMV reactivation and its viral load kinetics in critically ill patients with ANP

Objectives To study the prevalence of Cytomegalovirus (CMV) reactivation and its viral load kinetics in critically ill adult patients with acute necrotizing pancreatitis

Methodology Study design This prospective observational study will be conducted at the Department of Critical Care Medicine in collaboration with the Department of Gastroenterology and Microbiology, SGPGIMS, Lucknow after approval from the Institutional Ethics Committee (IEC).

Study protocol During the study period, all adult ICU patients with the diagnosis of acute necrotizing pancreatitis will be considered for inclusion. As per inclusion and exclusion criteria, these patients will be screened for the presence of Anti CMV IgG antibodies in their blood. If the patient is IgG seropositive and meets inclusion/exclusion criteria then they will be included in the study and followed up for CMV reactivation during their ICU stay. In patients having CMV reactivation, viral load kinetics will be further followed-up for the next 2 weeks.

Sample collection Blood samples: 1.0 ml blood will be collected in an EDTA vial from an existing venous catheter, on a weekly basis to find CMV reactivation during their ICU stay or 10th week of illness (whichever comes first).

Percutaneous drain: If the patient had an abdominal drain in the proximity of the pancreas, 2.0 ml will be collected in a sterile container on a weekly basis to find CMV reactivation during their ICU stay or the 10th week of illness (whichever comes first).

Pancreatic necrosum: If the patient underwent for necrosectomy, then pancreatic necrosum will be collected in a sterile container (single time)

Laboratory analysis ELISA for IgG antibody detection: The serum collected will be tested for IgG antibodies by ELISA as per manufacturer recommendations. (Abbott Laboratories, Abbott Park, IL). The cut-off of will be set at 0.5 WHO IU/ml (Calibrator 2) by the kit's manufacturer. Samples with a concentration higher than 0.5 WHO IU/ml will be considered positive for CMV IgG. All samples will be tested in duplicate.

CMV quantitative real-time PCR:

DNA Extraction: DNA extraction will be performed on 200 μl of a sample using a QIAamp DNA kit (Qiagen, Inc., Valencia, Calif.). Then, 60 μl of Tris (10 mM, pH 8.0) will be used to elute the DNA, and 10 μl of the DNA will be used for each PCR. The extracted DNA will be stored at -800 C for further work.

Quantitative Real-time PCR for virus detection: A 25 μL reaction will be prepared for the detection of CMV by RTPCR utilizing 10 μL of extracted DNA, 12.5 μL of 2X PCR buffer, and 1.5 μL of AgPath RT-PCR Reagents (Thermo Fisher Scientific, Massachusetts USA) and 1 μL Primer and probe sequences described elsewhere. All oligonucleotides will be synthesized and procured from Thermo Fisher Scientific, USA, and thermal cycling will be performed at 95 °C for 3 min and then 40 cycles of 95 °C for 15 s, 58 °C for the 30s using Applied bio system 7500 Real-Time PCR system (Thermo Fisher Scientific, Massachusetts USA). Each test will consist of 5 quantitative control and results will be interpreted accordingly.

Definitions Acute necrotizing pancreatitis: This will be diagnosed on the basis of clinical sign-symptoms / laboratory parameters and the presence of non-enhancing areas of the pancreas on a contrast-enhanced CT (CECT) scan.

CMV reactivation: The cut-off for diagnosing CMV reactivation will be taken as a value of >1000 copies/ml.

Data collections Demographic and relevant clinical characteristics of included patients will be collected on a structured case report form.

Sample size and statistical analysis Among screened acute necrotizing pancreatitis, 95% of patients are expected to have seropositive for IgG. Assuming 50% seropositive (IgG) patients will develop Cytomegalovirus (CMV) reactivation during the ICU stay. Taking a 15% margin of error in the assumed prevalence (i.e. expected range of 35 to 65%), at a two-sided 95% Confidence interval, the estimated sample size is 43. This study is time limited is 18 months and so during the study period all eligible patients will be screened and considered for inclusion in this study. The investigators are expecting about 50 patients.

Descriptive statistics of the continuous variables are to be presented as mean± standard deviation/median (inter-quartile range) while categorical variables in frequency (%) as appropriate. Student's t-test (independent as well as paired-samples t-test as appropriate) or its non-parametric methods to be used to compare the means/medians between the two groups whereas the Chi-square test or Fisher exact test will be used to compare the proportions. The incidences of CMV reactivations will be calculated and this association with demographic and clinical factors to be assessed using univariate as well as multivariate Cox proportional hazard models. A p-value < 0.05 will be considered statistically significant. Statistical package for social sciences, version-23 (SPSS-23, IBM, Chicago, USA), and MedCalc Software will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute necrotizing pancreatitis patients who require ICU admission, with at least a two-week duration of illness and the presence of CMV seropositivity (Anti CMV IgG antibodies).

Exclusion Criteria:

* Age < 18 years
* Expected survival < 72 hours
* Duration of pancreatitis more than 10 weeks
* Use of antiviral agents within the last 7 days
* Known or suspected underlying immune deficiency (history of solid organ or stem cell transplantation, infection with the human immunodeficiency virus, hematological malignancy, use of immunosuppressive medication (more than 0.1mg/kg prednisone for >3 months, more than 75mg/day prednisone for >3 weeks or equivalent), chemotherapy /radiotherapy in the year before ICU admission and any known humeral or cellular immune deficiency
* Pregnancy
* Patients who do not consent to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute necrotizing pancreatitis patients who require ICU admission
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Cytomegalovirus (CMV) reactivation in critically ill adult patients with acute necrotizing pancreatitis | From the date of inclusion in the study until the day of discharge from the ICU or up to 10 weeks of illness, whichever came first
  Percentage of included patients (CMV seropositive IgG) who had viral load >1000/cc
Cytomegalovirus (CMV) viral load kinetics in critically ill adult patients with acute necrotizing pancreatitis | From the date of CMV reactivation until 2 weeks thereafter or the day of discharge from the ICU, whichever came first
  Changes in CMV viral load count during their clinical course

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS); Atul Garg, MD, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Department of Critical Care Medicine, Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beger HG, Rau BM. Severe acute pancreatitis: Clinical course and management. World J Gastroenterol. 2007 Oct 14;13(38):5043-51. doi: 10.3748/wjg.v13.i38.5043. PMID 17876868
- [Background] Thoeni RF. The revised Atlanta classification of acute pancreatitis: its importance for the radiologist and its effect on treatment. Radiology. 2012 Mar;262(3):751-64. doi: 10.1148/radiol.11110947. PMID 22357880
- [Background] Beger HG, Rau B, Isenmann R. Natural history of necrotizing pancreatitis. Pancreatology. 2003;3(2):93-101. doi: 10.1159/000070076. No abstract available. PMID 12774801
- [Background] Banks PA, Freeman ML; Practice Parameters Committee of the American College of Gastroenterology. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006 Oct;101(10):2379-400. doi: 10.1111/j.1572-0241.2006.00856.x. No abstract available. PMID 17032204
- [Background] Frossard JL, Steer ML, Pastor CM. Acute pancreatitis. Lancet. 2008 Jan 12;371(9607):143-52. doi: 10.1016/S0140-6736(08)60107-5. PMID 18191686
- [Background] Petrov MS, Shanbhag S, Chakraborty M, Phillips AR, Windsor JA. Organ failure and infection of pancreatic necrosis as determinants of mortality in patients with acute pancreatitis. Gastroenterology. 2010 Sep;139(3):813-20. doi: 10.1053/j.gastro.2010.06.010. Epub 2010 Jun 9. PMID 20540942
- [Background] Reber HA. Pathogenesis of infection in pancreatic inflammatory disease. Pancreatology. 2001;1(3):207-9. doi: 10.1159/000055811. No abstract available. PMID 12120195
- [Background] Jain S, Mahapatra SJ, Gupta S, Shalimar, Garg PK. Infected Pancreatic Necrosis due to Multidrug-Resistant Organisms and Persistent Organ failure Predict Mortality in Acute Pancreatitis. Clin Transl Gastroenterol. 2018 Oct 5;9(10):190. doi: 10.1038/s41424-018-0056-x. PMID 30287818
- [Background] Trikudanathan G, Navaneethan U, Vege SS. Intra-abdominal fungal infections complicating acute pancreatitis: a review. Am J Gastroenterol. 2011 Jul;106(7):1188-92. doi: 10.1038/ajg.2010.497. PMID 21731015
- [Background] Schmidt PN, Roug S, Hansen EF, Knudsen JD, Novovic S. Spectrum of microorganisms in infected walled-off pancreatic necrosis - impact on organ failure and mortality. Pancreatology. 2014 Nov-Dec;14(6):444-9. doi: 10.1016/j.pan.2014.09.001. Epub 2014 Sep 16. PMID 25266641
- [Background] Moka P, Goswami P, Kapil A, Xess I, Sreenivas V, Saraya A. Impact of Antibiotic-Resistant Bacterial and Fungal Infections in Outcome of Acute Pancreatitis. Pancreas. 2018 Apr;47(4):489-494. doi: 10.1097/MPA.0000000000001019. PMID 29517630
- [Background] Reuken PA, Albig H, Rodel J, Hocke M, Will U, Stallmach A, Bruns T. Fungal Infections in Patients With Infected Pancreatic Necrosis and Pseudocysts: Risk Factors and Outcome. Pancreas. 2018 Jan;47(1):92-98. doi: 10.1097/MPA.0000000000000965. PMID 29215543
- [Background] Rasch S, Mayr U, Phillip V, Schmid RM, Huber W, Algul H, Lahmer T. Increased risk of candidemia in patients with necrotising pancreatitis infected with candida species. Pancreatology. 2018 Sep;18(6):630-634. doi: 10.1016/j.pan.2018.07.005. Epub 2018 Jul 14. PMID 30017450
- [Background] Werge M, Roug S, Novovic S, Schmidt PN, Hansen EF, Knudsen JD. Fungal Infections in Patients With Walled-off Pancreatic Necrosis. Pancreas. 2016 Nov;45(10):1447-1451. doi: 10.1097/MPA.0000000000000675. PMID 27518465
- [Background] Papazian L, Hraiech S, Lehingue S, Roch A, Chiche L, Wiramus S, Forel JM. Cytomegalovirus reactivation in ICU patients. Intensive Care Med. 2016 Jan;42(1):28-37. doi: 10.1007/s00134-015-4066-9. Epub 2015 Sep 30. PMID 26424680
- [Background] Docke WD, Prosch S, Fietze E, Kimel V, Zuckermann H, Klug C, Syrbe U, Kruger DH, von Baehr R, Volk HD. Cytomegalovirus reactivation and tumour necrosis factor. Lancet. 1994 Jan 29;343(8892):268-9. doi: 10.1016/s0140-6736(94)91116-9. PMID 7905100
- [Background] Kutza AS, Muhl E, Hackstein H, Kirchner H, Bein G. High incidence of active cytomegalovirus infection among septic patients. Clin Infect Dis. 1998 May;26(5):1076-82. doi: 10.1086/520307. PMID 9597229
- [Background] Cook CH, Trgovcich J, Zimmerman PD, Zhang Y, Sedmak DD. Lipopolysaccharide, tumor necrosis factor alpha, or interleukin-1beta triggers reactivation of latent cytomegalovirus in immunocompetent mice. J Virol. 2006 Sep;80(18):9151-8. doi: 10.1128/JVI.00216-06. PMID 16940526
- [Background] Hummel M, Abecassis MM. A model for reactivation of CMV from latency. J Clin Virol. 2002 Aug;25 Suppl 2:S123-36. doi: 10.1016/s1386-6532(02)00088-4. PMID 12361763
- [Background] Clari MA, Aguilar G, Benet I, Belda J, Gimenez E, Bravo D, Carbonell JA, Henao L, Navarro D. Evaluation of cytomegalovirus (CMV)-specific T-cell immunity for the assessment of the risk of active CMV infection in non-immunosuppressed surgical and trauma intensive care unit patients. J Med Virol. 2013 Oct;85(10):1802-10. doi: 10.1002/jmv.23621. Epub 2013 Jul 19. PMID 23868746
- [Background] Venet F, Davin F, Guignant C, Larue A, Cazalis MA, Darbon R, Allombert C, Mougin B, Malcus C, Poitevin-Later F, Lepape A, Monneret G. Early assessment of leukocyte alterations at diagnosis of septic shock. Shock. 2010 Oct;34(4):358-63. doi: 10.1097/SHK.0b013e3181dc0977. PMID 20220566
- [Background] Ziemann M, Sedemund-Adib B, Reiland P, Schmucker P, Hennig H. Increased mortality in long-term intensive care patients with active cytomegalovirus infection. Crit Care Med. 2008 Dec;36(12):3145-50. doi: 10.1097/CCM.0b013e31818f3fc4. PMID 18936696
- [Background] Jaber S, Chanques G, Borry J, Souche B, Verdier R, Perrigault PF, Eledjam JJ. Cytomegalovirus infection in critically ill patients: associated factors and consequences. Chest. 2005 Jan;127(1):233-41. doi: 10.1378/chest.127.1.233. PMID 15653989
- [Background] Limaye AP, Kirby KA, Rubenfeld GD, Leisenring WM, Bulger EM, Neff MJ, Gibran NS, Huang ML, Santo Hayes TK, Corey L, Boeckh M. Cytomegalovirus reactivation in critically ill immunocompetent patients. JAMA. 2008 Jul 23;300(4):413-22. doi: 10.1001/jama.300.4.413. PMID 18647984
- [Background] Osawa R, Singh N. Cytomegalovirus infection in critically ill patients: a systematic review. Crit Care. 2009;13(3):R68. doi: 10.1186/cc7875. Epub 2009 May 14. PMID 19442306
- [Background] Lachance P, Chen J, Featherstone R, Sligl WI. Association Between Cytomegalovirus Reactivation and Clinical Outcomes in Immunocompetent Critically Ill Patients: A Systematic Review and Meta-Analysis. Open Forum Infect Dis. 2017 Feb 13;4(2):ofx029. doi: 10.1093/ofid/ofx029. eCollection 2017 Spring. PMID 29497626
- [Background] Li X, Huang Y, Xu Z, Zhang R, Liu X, Li Y, Mao P. Cytomegalovirus infection and outcome in immunocompetent patients in the intensive care unit: a systematic review and meta-analysis. BMC Infect Dis. 2018 Jun 28;18(1):289. doi: 10.1186/s12879-018-3195-5. PMID 29954328
- [Background] Ong DSY, Spitoni C, Klein Klouwenberg PMC, Verduyn Lunel FM, Frencken JF, Schultz MJ, van der Poll T, Kesecioglu J, Bonten MJM, Cremer OL. Cytomegalovirus reactivation and mortality in patients with acute respiratory distress syndrome. Intensive Care Med. 2016 Mar;42(3):333-341. doi: 10.1007/s00134-015-4071-z. Epub 2015 Sep 28. PMID 26415682
- [Background] Ong DSY, Bonten MJM, Spitoni C, Verduyn Lunel FM, Frencken JF, Horn J, Schultz MJ, van der Poll T, Klein Klouwenberg PMC, Cremer OL; Molecular Diagnosis and Risk Stratification of Sepsis Consortium. Epidemiology of Multiple Herpes Viremia in Previously Immunocompetent Patients With Septic Shock. Clin Infect Dis. 2017 May 1;64(9):1204-1210. doi: 10.1093/cid/cix120. PMID 28158551
- [Derived] Singh U, Gurjar M, Garg A, Mohindra S, Mishra P, Rahul R, Yadav SS, Azim A, Poddar B. Cytomegalovirus Reactivation in Critically Ill Patients With Acute Necrotizing Pancreatitis. Open Forum Infect Dis. 2025 Jul 23;12(8):ofaf438. doi: 10.1093/ofid/ofaf438. eCollection 2025 Aug. PMID 40838259